CLINICAL TRIAL: NCT06738511
Title: Validation of a Molecular Signature for Early Detection of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ADVANCED MARKER DISCOVERY S.L. (Industry)
Collaborators: European Union H2020 SME Instrument (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AMD-EUC-2016
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Screening; Advanced Adenomas (AA)
Keywords: colon and rectum cancer; in vitro diagnostic; liquid biopsy; screening programme
MeSH Terms: conditions — Rectal Neoplasms | interventions — Blood Specimen Collection; Colonoscopy

STUDY DESIGN:
Masking Description: Laboratory Technicians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood and Stool sampling (Other): To collect blood sampling (by the medical staff) and stool sampling (by the participant)
  Interventions: Diagnostic Test: blood sampling; Other: stool sampling; Other: colonoscopy

INTERVENTIONS:
Diagnostic Test: blood sampling — Molecular signature using plasma sample
Other: stool sampling — Stool sampling (by the participant)
Other: colonoscopy — Colonoscopy will be performed in the course of a screening programme

SUMMARY:
The goal of this Multicentre and international prospective study is to validate a molecular signature using plasma samples in average-risk population for colorectal cancer who undergo colonoscopy in a screening setting.

The main question it aims to answer is:

Does molecular signature in plasma sample have higher diagnostic accuracy than FIT for early detection of colorectal cancer? Participants who already have a colonoscopy as part of their regular medical care for colorectal cancer screening will provide a stool sample and a plasma sample.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 50 and 75 (both included) at the time of informed consent signed. They must understand the nature, significance, implications and risks of the clinical trial and must sign the informed consent form.
* Participants referred to the gastroenterology service who are going to undertake colonoscopy as a regular procedure for screening setting.
* Participants asymptomatic, average risk for CRC. Average risk is defined as those individuals who are age 50 or older with no history of adenoma, colorectal cancer, or inflammatory bowel disease, and with no family history of CRC (first degree relatives).

Exclusion Criteria:

* Participants between the ages of 50 and 75 (both included) at the time of Informed consent signature. They must understand the nature, significance, implications and risks of the clinical trial and must sign the informed consent form.
* Participants who have been diagnosed with CRC. The diagnosis must be subsequently confirmed by biopsy or surgery and pathological anatomy analysis during the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3421 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Demonstrate the diagnosis capacity of molecular signature in plasma samples | 48 months

SECONDARY OUTCOMES:
Demonstrate superiority of molecular signature in plasma samples compared with FIT | 48 months

OTHER OUTCOMES:
Performance of molecular signature in plasma samples (Diagnostic capability) in cases of false positive or false negatives obtained in FIT | 48 months

CONTACTS AND LOCATIONS:
Locations (2):
- MVZ für Gastroenterolgie am Bayerischen Platz, Berlin, Germany, Germany
- Narodowy Instytut Onkologii w Warszawie Zakład Profilaktyki Nowotworów, Warsaw, Poland, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quintero E, Castells A, Bujanda L, Cubiella J, Salas D, Lanas A, Andreu M, Carballo F, Morillas JD, Hernandez C, Jover R, Montalvo I, Arenas J, Laredo E, Hernandez V, Iglesias F, Cid E, Zubizarreta R, Sala T, Ponce M, Andres M, Teruel G, Peris A, Roncales MP, Polo-Tomas M, Bessa X, Ferrer-Armengou O, Grau J, Serradesanferm A, Ono A, Cruzado J, Perez-Riquelme F, Alonso-Abreu I, de la Vega-Prieto M, Reyes-Melian JM, Cacho G, Diaz-Tasende J, Herreros-de-Tejada A, Poves C, Santander C, Gonzalez-Navarro A; COLONPREV Study Investigators. Colonoscopy versus fecal immunochemical testing in colorectal-cancer screening. N Engl J Med. 2012 Feb 23;366(8):697-706. doi: 10.1056/NEJMoa1108895. PMID 22356323
- [Background] Lieberman D. Colonoscopy: as good as gold? Ann Intern Med. 2004 Sep 7;141(5):401-3. doi: 10.7326/0003-4819-141-5-200409070-00018. No abstract available. PMID 15353432
- [Background] Siegel and Jemal. American Cancer Society. Colorectal Cancer Facts & Figures 2011-2013. Atlanta: American Cancer Society, 2011.
- [Background] von Karsa L, Patnick J, Segnan N. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Executive summary. Endoscopy. 2012 Sep;44 Suppl 3:SE1-8. doi: 10.1055/s-0032-1309822. Epub 2012 Sep 25. PMID 23012113